CLINICAL TRIAL: NCT05557877
Title: Targeted Prevention of Postpartum-Related Breast Cancer
Brief Title: Low Dose Aspirin for the Prevention of Postpartum Related Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MC220301; R01CA262393 (NIH); NCI-2022-07430 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC220301 (Other: Mayo Clinic); 22-000606 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling; Aspirin; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (low-dose aspirin) (Experimental): Patients undergo standard of care breast biopsy for assessment of abnormalities seen on imaging, as well as collection of blood during screening. If cancer is found, patient is taken off study and treatment options are discussed with treating physician.
  Patients without a cancer finding on biopsy then receive low-dose aspirin by mouth daily for 42-65 days and undergo collection of blood on study. Patients may undergo breast biopsy as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Drug: Low-Dose Aspirin; Other: Questionnaire Administration; Procedure: Biopsy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Low-Dose Aspirin — Given PO
  Other Names: Baby Aspirin
Other: Questionnaire Administration — Ancillary studies
Procedure: Biopsy — Undergo breast biopsy
  Other Names: Bx

SUMMARY:
This phase II trial tests whether low-dose aspirin can affect markers of inflammation in postpartum (after childbirth) women planning to have a breast biopsy. Chronic inflammation may increase the risk of postpartum related breast cancer. Low-dose aspirin is a non-steroidal anti-inflammatory drug. Giving low-dose aspirin may affect markers of inflammation in blood and tissue and may prevent postpartum related breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Pre- versus (vs.) post-intervention change in post-partum-related breast cancer (PRBC) score.

SECONDARY OBJECTIVE:

I. Pre- vs. post-intervention change in postpartum involution (PPI) signature score.

EXPLORATORY OBJECTIVES:

I. Pre- vs. post-intervention change in percent of epithelial cells positive for COX-2, estrogen receptor (ER)/Ki67, gammaH2AX, and p16 in "normal" and in benign breast disease (BBD) lobule.

II. Pre- vs. post-intervention change in serum C-reactive protein (CRP), estrogens, insulin/insulin-like growth factors (IGFs), and adipokines.

III. Pre- vs. post-intervention changes in tissue and urine prostaglandins (PGs) and PGE2.

OUTLINE:

Patients undergo standard of care breast biopsy for assessment of abnormalities seen on imaging, as well as collection of blood during screening. If cancer is found, patient is taken off study and treatment options are discussed with treating physician.

Patients without a cancer finding on biopsy then receive low-dose aspirin orally (PO) daily and undergo collection of blood on study. Patients may undergo breast biopsy as clinically indicated.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Age >= 18 years and =< 45 years of age
* PRE-REGISTRATION: Willingness to provide mandatory tissue specimens for correlative research at two timepoints.
* PRE-REGISTRATION: Had a live birth =< 10 years prior to pre-registration
* PRE-REGISTRATION: Pre-menopausal according to patient report and/or clinical determination
* PRE-REGISTRATION: Provide written informed consent
* PRE-REGISTRATION: Ability to complete questionnaire(s) by themselves or with assistance
* PRE-REGISTRATION: Willingness to provide mandatory blood and urine specimens for correlative research
* REGISTRATION: Age >= 18 years and =< 45 years of age
* REGISTRATION: Registration for this study must be completed either =< one (1) year after the qualifying pre-registration biopsy is performed for this study or =< one (1) year after collection of the archived tissue (for those who did not have a pre-registration biopsy performed after pre-registration for this study)
* REGISTRATION: Hemoglobin >= 9.0 g/dL (obtained =< 30 days prior to registration)
* REGISTRATION: Platelet count >= 100,000/mm^3 (obtained =< 30 days prior to registration
* REGISTRATION: Serum creatinine =< 2.0 mg/dl (obtained =< days prior to registration)
* REGISTRATION: Negative pregnancy test done =< 14 days prior to registration
* REGISTRATION: Willing to use contraception while on treatment
* REGISTRATION: Provide written informed consent
* REGISTRATION: Ability to complete questionnaire(s) by themselves or with assistance
* REGISTRATION: Willingness to provide mandatory blood and urine specimens for correlative research
* REGISTRATION: Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* PRE-REGISTRATION: History of breast cancer including ductal breast carcinoma in situ (DCIS)
* PRE-REGISTRATION: Received systemic treatment for any other cancer at any time
* PRE-REGISTRATION: Currently taking aspirin or other non-steroidal anti-inflammatory drugs (NSAIDS) (no doses within =< 5 days prior to pre-registration and no more than four doses within =< 30 days prior to pre-registration)
* PRE-REGISTRATION: Currently taking other agents for the prevention of breast cancer
* PRE-REGISTRATION: Currently taking anticoagulants
* PRE-REGISTRATION: Contraindication for aspirin use
* PRE-REGISTRATION: Known or suspected active breast infection
* REGISTRATION: Known DCIS or invasive cancer
* REGISTRATION: No research tissue available from pre-registration biopsy or from archived tissue (collected =< 12 months prior to pre-registration)
* REGISTRATION: Currently taking aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs) (NOTE: no doses within =< 5 days prior to registration and no more than four doses within =< 30 days prior to registration)
* REGISTRATION: Co-morbid illnesses/conditions which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* REGISTRATION: Any contraindication to aspirin use including but not limited to:

  * Bleeding disorders (e.g., hemophilia)
  * Stomach or intestinal bleeding =< 6 months prior to registration
  * Known allergy to other non-steroidal anti-inflammatory drugs (NSAIDs)
* REGISTRATION: Currently taking anticoagulants
* REGISTRATION: Any prior or current malignancy requiring prior or current systemic therapy
* REGISTRATION: Currently pregnant or planning to become pregnant in the next 90 days
* REGISTRATION: Post-menopausal:

  * Prior bilateral surgical oophorectomy or
  * No menses for > 1 year with estradiol levels within postmenopausal range, according to institutional standard
* REGISTRATION: Known or suspected active breast infection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in pregnancy-related breast cancer (PRBC) score | Up to 30 days
  Assessed using pre- versus post-treatment PRBC scores. Patients who are eligible, consented, received at least 70% of the study treatment, and provided both a pre- and post-intervention tissue specimen will be evaluated for this outcome.

SECONDARY OUTCOMES:
Change in postpartum involution (PPI) signature score | Up to 30 days
  Assessed using pre- and post-intervention PPI signature scores for each person.

OTHER OUTCOMES:
Change in percent of epithelial cells positive for COX-2, estrogen receptor (ER)/Ki67, gammaH2AX, and p16 in "normal" and in benign breast disease (BBD) lobules | Up to 30 days
  The change in percent of positive epithelial pre- and post-intervention will be assessed for each person.
Change in serum C-reactive protein (CRP), estrogens, insulin/insulin-like growth factors (IGFs), and adipokines | Up to 30 days
  Serum values will be measured pre- and post-intervention for each person.
Changes in tissue and urine prostaglandins (PGs) and PGE2 | Up to 30 days
  PGs will be measured pre- and post-intervention for each person.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn J. Ruddy, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Indiana University Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials